CLINICAL TRIAL: NCT01424657
Title: Magnetic Resonance Cholangiopancreatography Versus Endoscopic Retrograde Cholangiopancreatography in the Approach to Patients With Suspected Biliary Obstruction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated before reaching the estimated sample size because of trial fatigue.
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Alberta Heritage Foundation for Medical Research (Other); American College of Gastroenterology (Other); American Digestive Health Foundation (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Alan Barkun, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC. 97-026
Record Dates: First submitted 2011-08-23; First posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Suspected Biliary Obstruction
Keywords: MRCP; ERCP; BILIARY OBSTRUCTION; EFFECTIVENESS
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ERCP (Experimental): ERCP is an endoscopic examination that allows opacification of the biliary tree by direct injection into the common bile duct through its distal opening in the duodenum at the ampulla of Vater
  Interventions: Procedure: ERCP
- MRCP (Experimental): The magnetic resonance cholangiopancreatography (MRCP)allows direct visualization of the biliary tree and pancreatic duct, similar to contrast cholangiography, but without the need for administration of contrast medium
  Interventions: Procedure: MRCP

INTERVENTIONS:
Procedure: ERCP — Endoscopic retrograde cholangiopancreatography
  Arms: ERCP
Procedure: MRCP — magnetic resonance cholangiopancreatography
  Arms: MRCP

SUMMARY:
The main objective of this study is to assess the effectiveness and costs of magnetic resonance cholangiopancreatography (MRCP) and compare it to endoscopic retrograde cholangiopancreatography (ERCP) in the work up of patients with suspected bile duct obstruction on ultrasound. The investigators do not anticipate that a universal recommendation for a given diagnostic test (MRCP versus ERCP) will be applicable in all patients presenting with bile duct obstruction. Rather, the investigators hope to provide quantitative and comparative data relevant to the different clinical situations likely to be encountered in practice, in order to assist physicians in choosing the appropriate diagnostic modality. More specifically, the investigators feel that patients with intrahepatic or hilar obstruction (particularly those with malignant conditions), and those with partial common bile duct (CBD) obstruction (to rule out suspected choledocholithiasis) will benefit most from this new technology and the avoidance of an unnecessary ERCP to further determine the biliary anatomy.

DETAILED DESCRIPTION:
The approach to investigation and management of intermediate-risk biliary obstruction is controversial. Both magnetic resonance cholangiopancreatography(MRCP)and endoscopic retrograde cholangiopancreatography (ERCP) are used interchangeably in practice, with little literature to support the efficacy of one versus the other.

The purpose is to assess the effectiveness of MRCP compared to ERCP in the initial work-up of patients at intermediate risk of suspected biliary obstruction following initial clinical assessment and ultrasonography.

A randomized medical effectiveness study was conducted across three tertiary care hospital sites. Patients at intermediate risk of biliary obstruction were randomized to either ERCP or MRCP based on level of obstruction as seen by ultrasound (US).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Elevated bilirubin (>30 umol/L)
* CBD dilatation on ultrasound: greater than 7 mm wide with gallbladder in situ, or 10mm wide in patient post-cholecystectomy
* Suspected or detected gallstone on ultrasound

Exclusion Criteria:

* Low probability of biliary tract disease
* Active cholangitis
* Bilio-pancreatic pathology identified on ultrasound or CT scan
* Any clinical condition precluding MRCP or ERCP: severe cardio-respiratory disease, pregnancy, significant coagulopathy (INR over 1.5)
* Presence of Roux-en-Y bilio-enteric anastomosis
* Any metallic implant making ERCP or MRCP hazardous
* ERCP or MRCP performed within 6 months prior to study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 1997-10; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
occurrence of adverse biliary events | 12 months
  The goal of this study was to evaluate the effectiveness of MRCP compared to ERCP in assessment of patients at intermediate risk for suspected biliary obstruction

SECONDARY OUTCOMES:
complication-related length of stay | 12 months
Number of additional procedures (i.e ERCP, MRCP, US...) | 12 months
mortality | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- MUHC- McGill University Health Center, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Bhat M, Romagnuolo J, da Silveira E, Reinhold C, Valois E, Martel M, Barkun JS, Barkun AN. Randomised clinical trial: MRCP-first vs. ERCP-first approach in patients with suspected biliary obstruction due to bile duct stones. Aliment Pharmacol Ther. 2013 Nov;38(9):1045-53. doi: 10.1111/apt.12481. Epub 2013 Sep 11. PMID 24024705